CLINICAL TRIAL: NCT07268222
Title: Metyrapone Versus Osilodrostat in Patients With Metabolic Autonomous Cortisol Secretion (MACS)
Acronym: MOMACS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Anna Angelousi, associate professor, Laikο General Hospital, Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Laikon
Record Dates: First submitted 2025-11-21; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Mild Autonomous Cortisol Secretion (MACS)
Keywords: cortisol; Cushing; MACS; METYRAPONE; osilodrostat
MeSH Terms: interventions — Metyrapone; Osilodrostat; Surgical Procedures, Operative; Adrenalectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with MACS (Other): Patients with MACS (Adults > 18 years old with 1mg ODST F levels >1.8μg/dl and normal or slightly abnormal UFC OR midnight salivary cortisol levels AND no symptoms or signs of overt hypercortisolism.)
  Interventions: Drug: Metyrapone 250 mg Oral Tablets; Drug: Osilodrostat 1 MG; Procedure: adrenalectomy; Other: Watch and wait

INTERVENTIONS:
Drug: Metyrapone 250 mg Oral Tablets — metyrapone( 250 -750 mg) vs. osilodrostat (1-3 mg) vs. surgery vs watch and wait strategy in the management of patients with MACS
  Other Names: osilodrostat; surgery
Drug: Osilodrostat 1 MG — administration of 1-3 mg of osilodrostat at 19.00
Procedure: adrenalectomy — Surgery performed in patients with MACS
Other: Watch and wait — Follow-up

SUMMARY:
This study will compare the efficacy and safety of the two 11β-hydroxylase inhibitors-metyrapone and osilodrostat-in patients with MACS.

Primary outcome To compare the efficacy (biochemical and clinical) of the two 11β-hydroxylase inhibitors (CYP11B1), metyrapone and osilodrostat, in patients with MACS not treated surgically (mainly bilateral adenomas or adrenal hyperplasias), as well as their side effects at time 0-, 3- and 6-months post-treatment.

Secondary outcome To evaluate alterations in clinical parameters (Blood Pressure, Body Mass Index-BMI), metabolic parameters (fasting blood glucose, insulin, Hb1Ac, HOMA, OGTT and lipids levels) at time 0-, 3- and 6-month after the initiation of the treatment and their effect on Bone Mineral Density (BMD) 1 year post-diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old with MACS and unilateral or bilateral adrenal adenomas or hyperplasia (based on imaging)
* 1 mg overnight dexamethasone suppression test (ODST): Cortisol levels at 8.00 am>1.8 μg/dl AND i) ACTH< 15 pg/ml OR ii) abnormal midnight salivary cortisol OR iii) Urinary free cortisol levels (UFC) /24h ≥ of the UNL

Exclusion Criteria:

* Abnormal liver enzymes
* eGFR < 40 ml/min/1.73 m3
* Pseudocushing syndrome
* Patients with any malignancy (active or past history), including ACC
* ACTH-dependent Cushing syndrome (Cushing disease or ectopic Cushing syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Comparison of the efficacy of metyrapone and osilodrostat | Baseline ( at t=0), at t=3 months and at =6 months
  Blood tests measuring baseline moring cortisol (μg/dl) levels pre and post-treatment
Comparison of the efficacy of metyrapone and osilodristat | Baseline (at t= 0), at t= 3 months and t= 6 months
  Measurement of the baseline morning ACTH (pg/ml) pre and post-treatment
Comparison of the efficacy of metyrapone and osilodristat | Baseline ( at t=0), at t=3 months and at t=6 months
  Measurement of the baseline morning DHEAS levels (μg/dl) pre and post-treatment
Comparison of the efficacy of metyrapone and osilodristat | Baseline ( at t=0), at t=3 months and at =6 months
  Measurement of urinary free cortisol (μg/24h) pre and post-treatment
Comparison of metyrapone and osilodrostat efficacy | Baseline (at t=0), at t=3 months , at t =6 months
  Measurement of salivary midnight cortisol (μg/dl) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0), at t= 3months, at t=6 months
  Alteartions of LDL levels (mg/dl) pre and post-treatment

SECONDARY OUTCOMES:
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline at t=0 , at 3 months and at 6 months
  Alterations of fasting blood glucose levels (mg/dl) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0), at t=3 months and at t=6 months
  Alteration of insuline levels (μU/ml) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0), at t=3 months and at t=6 months
  Alterations of Hb1Ac levels (%) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0) at t=3 months and t=6 months
  Alterations of HOMA-IR (glucose levels mmol/l x insuline levels mIU/L/22.5) pre and post -treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0), at t=3 months and at t=6 months
  Alterations of cholesterol levels (mg/dl) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0), at t=3 months and at t=6 months
  Alterations of triglycerides levels (mg/dl) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline (t=0), at t=3 months and at t=6 months
  Alterations of HDL levels (mg/dl) pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of alterations of metabolic parameters | Baseline at t=0, at t=3 months , at t=6 months
  Alterations of glucose levels post-OGTT pre and post-treatment

OTHER OUTCOMES:
Comparison of metyrapone and osilodrostat in terms of other parameters | Baseline (t=0), at t=3 months and t=6 months
  Alterations of systolic and diastolic blood pressure (mmHg) at morning pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of other parameters | Baseline (t=0), t=3 months , t=6 months
  Alterations of BMI (weight (kg) / height(cm2)) levels pre and post-treatment
Comparison of metyrapone and osilodrostat in terms of other parameters | Baseline at t=0 and at t= 1 year
  Alterations of bone mineral density (BMD) in gr /cm3 pre and post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Laikon General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No